CLINICAL TRIAL: NCT04774835
Title: Implementing Assisted Partner Services for HIV Testing and Treatment in Western Kenya
Brief Title: Assisted Partner Services and HIVST in Western Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Kenyatta National Hospital (Other Government); University of Nairobi (Other)
Responsible Party: Principal Investigator, Carey Farquhar, Professor, School of Medicine: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00002420; R01AI134130 (NIH)
Record Dates: First submitted 2021-02-14; First posted 2021-03-01 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Hiv
Keywords: HIV self-testing; Assisted partner services; Acceptability; Implementation Science
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard aPS (Active Comparator): Subjects receive standard assisted partner services from their local HIV testing services (HTS) counselor.
  Interventions: Diagnostic Test: Standard aPS
- aPS + HIVST (Experimental): Subjects receive standard assisted partner services from their local HIV testing services (HTS) counselor as well as the option to do HIV self-testing (HIVST) instead of testing at the local HTS location.
  Interventions: Diagnostic Test: HIVST

INTERVENTIONS:
Diagnostic Test: HIVST — aPS will be offered to sexually active men and women who test HIV seropositive at the study sites by facility staff supported by aPS advisors. Those accepting aPS will be asked to provide names and contact information (phone numbers; home and work addresses) for their sexual partners, and these partners will be contacted, notified anonymously of the HIV exposure, and offered HIV self-testing by HTS counselors working at the facilities. Any partner who tests HIV seropositive will receive assistance linking to care and registering in an HIV comprehensive care clinic. They will also receive aPS so that their partners can be notified and HIV tested. Follow-up of index clients will continue after testing through HTS locations and all partners will be followed to determine HIV testing and treatment outcomes.
  Arms: aPS + HIVST
Diagnostic Test: Standard aPS — aPS will be offered to sexually active men and women who test HIV seropositive at the study sites by facility staff supported by aPS advisors. Those accepting aPS will be asked to provide names and contact information (phone numbers; home and work addresses) for their sexual partners, and these partners will be contacted, notified anonymously of the HIV exposure, and offered HIV testing at their local HTS location by HTS counselors working at the facilities. Any partner who tests HIV seropositive will receive assistance linking to care and registering in an HIV comprehensive care clinic. They will also receive aPS so that their partners can be notified and HIV tested. Follow-up of index clients will continue after testing through HTS locations and all partners will be followed to determine HIV testing and treatment outcomes.
  Arms: Standard aPS

SUMMARY:
This study includes different designs with Aim 1 being a cluster randomized controlled trial to investigate the use of HIV self-testing (HIVST) as a mode of HIV testing in Western Kenya in addition to the standard of care, assisted partner services (aPS). Aim 2 includes focus group discussions, in-depth interviews, semi-structured interviews, direct observation of facility infrastructure and clinic procedures, and data extraction from facility and county/national databases and expenditure reports to study acceptability, costs, and implementation aspects of HIVST within the aPS framework.

ELIGIBILITY:
Inclusion Criteria:

Aim 1:

* Men and women
* Tests HIV positive and is not in care or on treatment
* ≥18 years old
* Willing and able to provide informed consent
* Able to provide locator information for sexual partners

Aim 2:

* ≥18 years old
* Willing and able to provide informed consent

Exclusion Criteria:

Aim 1:

* Pregnancy
* Reports intimate partner violence during last month
* <18 years old

Aim 2:

• <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4941 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Number of participants testing for the first time | 1 year
  Identify if there's a difference between standard aPS and aPS+HIVST in the number of participants choosing to get HIV tested for the first time.
Number of newly diagnosed HIV-infected or known positive and not in care | 1 year
  Identify if there's a difference between standard aPS and aPS+HIVST in the number of participants newly being diagnosed with HIV after participation, or those known to be positive but not currently under care.
Linking a new positive or known positive not in care to a treatment center | 1 year
  Identify if there's a difference between standard aPS and aPS+HIVST in the number of participants that are linked to care at a treatment center.
Initiating ART, or re-initiating ART if previously lost to follow-up | 1 year
  Identify if there's a difference between standard aPS and aPS+HIVST in the number of participants that initiate (or re-initiate) ART.

SECONDARY OUTCOMES:
Difficulty of using the HIVST kit | 1 year
  Understand the ease of using HIV self-testing kits in this population and setting, via a survey question with a 4 point Likert scale ranging from "very easy" to "very "hard".
Difficulty of interpreting the HIVST results | 1 year
  Understand the readability of HIV self-testing results in this population and setting, via a survey question.

CONTACTS AND LOCATIONS:
Overall Officials: Carey Farquhar, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy Paladhi U, Katz DA, Otieno G, Hughes JP, Lagat H, Masyuko S, Sharma M, Macharia P, Bosire R, Mugambi M, Kariithi E, Farquhar C. Effectiveness of HIV self-testing when offered within assisted partner services in Western Kenya (APS-HIVST Study): a cluster randomized controlled trial. J Int AIDS Soc. 2024 Jul;27 Suppl 1(Suppl 1):e26298. doi: 10.1002/jia2.26298. PMID 38965976